CLINICAL TRIAL: NCT02243228
Title: A Prospective Study of Inhaling Granulocyte-macrophage Colony Stimulating Factor in Adult Patients With Mild-to-moderate Autoimmune Pulmonary Alveolar Proteinosis in China: a Randomized Open-label Study
Brief Title: Inhalation of Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) for Autoimmune Pulmonary Alveolar Proteinosis (PAP)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Kaifeng Xu, MD, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XT 01
Record Dates: First submitted 2014-09-14; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Autoimmune Pulmonary Alveolar Proteinosis
Keywords: granulocyte-macrophage colony stimulating factor(GM-CSF); Autoimmune pulmonary alveolar proteinosis (PAP)
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis, Acquired | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GM-CSF, nebulizer (Experimental): After the patients were randomly divided into two groups, they will be treated by GM-CSF (using nebulizer, 150ug bid) every other week for 6 months.
  Interventions: Drug: GM-CSF

INTERVENTIONS:
Drug: GM-CSF
  Other Names: HUABEI JIMUXIN

SUMMARY:
The purpose of the study is to evaluate if inhaled granulocyte-macrophage colony stimulating factor delay the increase in alveolar-arterial oxygen difference, compared to no treatment, for adult patients with mild-to-moderate autoimmune pulmonary alveolar proteinosis in China over a two-year period.

DETAILED DESCRIPTION:
Autoimmune pulmonary alveolar proteinosis (PAP, previously known as idiopathic PAP) is a rare interstitial lung disease elicited by the formation of autoantibodies which neutralize the activity of granulocyte-macrophage colony-stimulating factor (GM-CSF) which decreases macrophage clearance of surfactant.

Currently, the standard treatment strategy for PAP is whole lung lavage (WLL)，which is invasive and has limitations. Inhaled GM-CSF therapy became a new option for PAP patients not only because of its effectiveness and safety, but it is convenient way for patients who are reluctant to do operation as well. We are planning to prospectively evaluate if inhaled granulocyte-macrophage colony stimulating factor would delay the increase in alveolar-arterial oxygen difference (A-aDO2, which is the most sensitive factor in evaluating APAP5), compared to placebo, for patients with mild-to-moderate autoimmune pulmonary alveolar over a two-year period.

A total of 42 subjects with APAP who meet the inclusion criteria will be enrolled at Peking Union Medical College Hospital and Nanjing Drum Tower Hospital. After observe APAP patients for 3 months to rule out patients who resolved spontaneously, the participants will undergo randomization (by random number table)and stratified into two different groups by their DSS. Then they will be treated by GM-CSF (using nebulizer, 150ug bid) every other week or no treatment for 6 months, and will be followed on an outpatient basis at 2 weeks, and 1, 3, 6, 9, 12, 15, 18, 21 and 24 months after initiation of therapy.

ELIGIBILITY:
Accessible population:

Adult patients with mild-to-moderate autoimmune pulmonary alveolar and without spontaneous remission will be enrolled at Peking Union Medical College Hospital and Nanjing Drum Tower Hospital.

Inclusion Criteria:

* Adult autoimmune PAP subjects will be included: 1) a positive PAS stain from BALF or lung biopsy; 2) high level of serum anti-GM-CSF antibody (>2.39ug/ml, the cut-off point in our hospital); 3) age above 18 years old; 4) exclude hereditary and secondary PAP.
* Able to give written informed consent and comply with the requirements of the study.
* Patients are not eligible for the whole lung lavage (WLL), decided by clinicians.
* Eligibility for GM-CSF inhalation: 1) Disease severity score (DSS) is 1-3; 2) No treatment with GM-CSF therapy or WLLin the 3 months prior to enrollment. Definition of DSS2: 1, no symptom and PaO2>=70mmHg；2, PaO2>=70mmHg with symptoms；3, PaO2>=60 and <70mmHg; 4, PaO2>=50 and <60mmHg; 5, PaO2<50mmHg.

Exclusion Criteria:

* Patients will be observed for 3 months and all APAP patients who resolved spontaneously will be excluded from our study.
* PAP resulting from another condition (e.g. occupational exposure to silica, underlying HIV, respiratory infections, myeloproliferative disorder or leukaemia);
* A normal or low-titre serum anti-GM-CSF antibody (≤2.39ug/ml);
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies；
* Chronic lung disease associated with already existing respiratory failure (such as pulmonary emphysema or fibrosis);
* Other serious medical conditions which, in the opinion of the investigator, would make the patient unsuitable for the study.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
A-aDO2 difference | 2 years

SECONDARY OUTCOMES:
Time to relapse | up to 2 years
  The definition of relapse were as follow: 1) newly requirement for whole lung lavage (WLL); or 2) PAP associated death; or 3) a reduction in PaO2 of more than 10mmHg, or an increase in DA-aO2 of more than 10mmHg; or 4) a worsen chest HRCT.
FEV1 difference | 2 years
6 minutes walking distance difference | 2 years
Severe adverse event | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Feng Xu, M.D., Principal Investigator — Peking Union Medical College Hosptial
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Tian X, Yang Y, Chen L, Sui X, Xu W, Li X, Guo X, Liu L, Situ Y, Wang J, Zhao Y, Meng S, Song W, Xiao Y, Xu KF. Inhaled granulocyte-macrophage colony stimulating factor for mild-to-moderate autoimmune pulmonary alveolar proteinosis - a six month phase II randomized study with 24 months of follow-up. Orphanet J Rare Dis. 2020 Jul 2;15(1):174. doi: 10.1186/s13023-020-01450-4. PMID 32615994